CLINICAL TRIAL: NCT03112889
Title: A Phase II Pilot Study to Explore Treatment With Sodium Valproate in Adults With McArdle Disease (Glycogen Storage Disorder Type V, GSDV)
Brief Title: Sodium Valproate for GSDV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11/0090
Record Dates: First submitted 2015-08-11; First posted 2017-04-13 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Glycogen Storage Disease Type V; McArdle Disease
Keywords: McArdle Disease; McArdle's Disease; Glycogen Storage Disease Type V; GSDV; Sodium Valproate; Valproic Acid; Myophosphorylase Deficiency; Muscle Phosphorylase Deficiency; Glycogenosis; Glycogen Storage Disorder
MeSH Terms: conditions — Glycogen Storage Disease Type V; Glycogen Storage Disease | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sodium Valproate (Experimental): Subjects will receive sodium valproate modified release 20mg/kg/day (maximum dose 2.0g/day) administered orally once daily for six months.
  Interventions: Drug: Sodium Valproate

INTERVENTIONS:
Drug: Sodium Valproate — Subjects will receive sodium valproate modified release 20mg/kg/day (maximum dose 2.0g/day) administered orally once daily for six months.

SUMMARY:
McArdle disease is a metabolic myopathy characterised by the absence of glycogen phosphorylase in skeletal muscle. Sodium Valproate is part of a group of drugs known as histone deacetylase inhibitors, which have a direct effect on chromatin. Recently a drug trial in an animal model of McArdle disease showed that sodium valproate stimulated the expression of a different isoform of the missing enzyme in skeletal muscle.

A safety and feasibility study of sodium valproate in people with McArdle disease has been carried out in London (UK) and Copenhagen (DK) since January 2015. Participants will receive 20mg/Kg/day of sodium valproate for 6 months. The primary outcome measure is exercise performance assessed by cycle ergometry. Pre and post-treatment skeletal muscle biopsies will be performed to assess for glycogen phosphorylase. Together with blood analyses for safety. Additional functional exercise tests will be performed.

DETAILED DESCRIPTION:
McArdle disease (Glycogen storage disease type V, GSDV) is an inherited metabolic disorder of skeletal muscle. Affected patients are unable to perform strenuous exercise due to a congenital absence of the enzyme muscle glycogen phosphorylase, essential for glycogen metabolism. This enzyme deficiency results in the inability to mobilise muscle glycogen stores from muscle, required for energy during strenuous exercise. In affected people symptoms of fatigue and cramps occur within minutes of initiating any activity and during strenuous activity such as lifting heavy weights or walking uphill, if activity is continued despite severe cramping, a contracture occurs which leads to muscle damage (rhabdomyolysis), myoglobinuria (dark brown/black discolouration of urine) and, when severe, acute renal failure.

Currently no satisfactory treatment can be recommended other than aerobic exercise. Although most people with McArdle disease have complete absence of skeletal muscle phosphorylase, there are a small minority of patients who possess splice site mutations that enable production of very small amounts (1-2%) of functional enzyme. These people have a milder phenotype with less severe symptoms, and functional exercise assessments have shown better exercise capacity than typical patients with the condition. Findings from these atypical individuals suggest potential therapeutic agents might only need to produce very small amounts of enzyme for significant functional improvement. Furthermore, finding a therapeutic agent to 'switch on' expression of the foetal isoenzyme may be a potential therapeutic strategy. There is some evidence from animal studies to suggest that sodium valproate can 'switch on' the foetal phosphorylase isoenzyme. The current proposes to undertake a feasibility study of 8 participants recruited in the UK and 7 in Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects and post-menopausal or infertile females
* Diagnosed with GSDV and over 18 years of age
* Normal serum carnitine level and acylcarnitine blood profile at screening visit

Exclusion Criteria:

* Children under the age of 18 years
* People older than 64 years
* Females of child bearing potential
* Patients with Diabetes
* Inflammatory disorders especially systemic lupus erythematosis.
* A previous history of sensitivity/allergy to sodium valproate and its excipients
* Patients treated with sodium valproate for epilepsy or a psychiatric disorder within the last 12 months prior to screening
* Patients with pre-existing liver disease or a family history of severe liver disease affecting a first degree relative. Liver disease will be defined by abnormal liver biopsy. Patients with GSDV may have raised serum transaminases that originate from muscle but which may cause abnormal liver function tests measured in serum, this will not be a reason for exclusion.
* Patients prescribed other anti-convulsant medication or any other medication known to interact with sodium valproate (see section 9.3).
* Patients who are sensitive to local anaesthetics that would prevent muscle biopsy.
* Subjects with any co-morbid illness or disability which would prevent an exercise assessment such as severe unstable/ untreated ischaemic heart disease, lower limb disability such as severe muscle weakness with muscle strength assessed as worse than MRC scale 3 in any pelvic girdle muscle.
* Inability to exercise due to a lower limb fracture would be an exclusion criterion until there is complete recovery of the injury.
* Patients known to have porphyria or an affected first degree relative affected with porphyria will be excluded from the study.
* Patients known to have mitochondrial disease or where there is a first degree relative with mitochondrial disease.
* Patients with a history of abnormal acyl carnitine profile or low serum carnitine level
* Male participants unwilling to use contraception

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

PRIMARY OUTCOMES:
Change in VO2peak | Week 1, Week 16 and Week 28
  The aerobic power will be measured at peak workload after a +- 15 minutes incremental cycle test performed on a cycle ergometer after 15 minutes constant load cycling.

SECONDARY OUTCOMES:
Presence of phosphorylase positive fibres | Week 0 and Week 28
  Pre and post-treatment muscle biopsies will be evaluated for phosphorylase enzyme activity
Change in total walked distance | Week 1, Week 16 and Week 28
  The total walked distance will be measured by the 12 minute walk test (corridor).
Blood lactate responses to exercise | Week 1, Week 16 and Week 28
  Lactate will be measured at rest, during a non-ischameic forearm exercise test (0, 2 and 5 minutes post exercise) and during a cycle test (5, 10 and 15 minutes during exercise and at exhaustion).
Safety of sodium valproate assessed by blood exams and self-reported adverse events | For the duration of the trial and within 3 months of Visit 3 (+- Week 40)
Adverse events log | Week 4, Week 8, Week 16, Week 20, Week 24, Week 28, +- Week 40
  Assessed during each study visit, monthly phone calls and symptoms diary
Quality of life | Week 1, Week 16 and Week 28
  Total score on SF36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ros Quinlivan, FRCPCH, MD, Principal Investigator — University College, London
Locations (2):
- Rigshospitalet, Copenhagen, Denmark
- MRC Centre for Neuromuscular Diseases, London, United Kingdom

REFERENCES:
- [Background] Howell JM, Dunton E, Creed KE, Quinlivan R, Sewry C. Investigating sodium valproate as a treatment for McArdle disease in sheep. Neuromuscul Disord. 2015 Feb;25(2):111-9. doi: 10.1016/j.nmd.2014.10.002. Epub 2014 Oct 13. PMID 25455802